CLINICAL TRIAL: NCT02443428
Title: Eribulin (HALAVEN) Use for the Treatment of Advanced Breast Cancer: A Prospective Observational Registry
Brief Title: Eribulin Use for the Treatment of Advanced Breast Cancer: A Prospective Observational Registry
Status: Completed | Type: Observational
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: OBU-N-H-01
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eribulin Mesilate: Participants will be treated in accordance with normal clinical practice. The recommend dose of eribulin is 1.23 mg/m2 administered intravenously on days 1 and 8 of every 21-day cycle. Treatment with eribulin is continued until disease progression, onset of unacceptable drug toxicities, or participant/physician's request to discontinue.

SUMMARY:
The purpose of this prospective observational registry is to monitor safety of eribulin in routine clinical practice. Additionally, this study will also assess the effectiveness of eribulin in real-life settings.

ELIGIBILITY:
Inclusion Criteria

The participants have to meet all of the following criteria to be eligible to enter into the prospective registry:

1. Participants older than 18 years of age
2. Willing and able to provide informed consent
3. Diagnosis of locally advanced or metastatic breast cancer
4. Progression after up to two previous chemotherapy regimens for advanced disease. Prior therapy should have included an anthracycline and a taxanes in either the adjuvant or advanced setting unless not suitable
5. Adequate bone marrow, liver, and renal function
6. Life expectancy greater than 12 weeks

Exclusion Criteria

Participants meeting the following criteria will not be permitted to enter the study:

1. Prior treatment with eribulin
2. Participants who have received more than two prior chemotherapeutic regimens for advanced disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with locally advanced or metastatic breast cancer who have progressed after up to two chemotherapeutic regimens for advanced disease will be prospectively included in the registry. Prior therapy should have included an anthracycline and a taxanes unless the patient was not suitable for these treatments.
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | From date of first administration of study drug up to 30 days after last administration of study drug or until approximately 2 years
  Safety assessment will consist of monitoring of all AEs, including SAEs at every visit. All participants will be evaluable for safety from the time of their first treatment with eribulin.

SECONDARY OUTCOMES:
Tumour response | From date of enrollment, Day 1 and Day 8 of every 21 day cycle or up to approximately 2 years
Overall survival (OS) | From date of first administration of study drug to date of death or up to approximately 2 years
Demographic and clinical characteristics | Up to approximately 2 years
Duration of treatment | Historical data collected at Baseline
Incidence of dose delays | From date of first administration up to approximately 2 years
Incidence of dose reductions | From date of first administration up to approximately 2 years
Relative dose intensity (RDI) of eribulin | From date of first administration up to approximately 2 years
Treatment patterns for locally advanced or metastatic breast cancer | Historical data collected at Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Kristeleit, Study Director — Guy's Hospital, Great Maze Pond
Locations (12):
- Denmark (2):
  - Aarhus
  - Copenhagen
- Dublin, Ireland
- United Kingdom (9):
  - Bath
  - Cottingham
  - Derby
  - London
  - Maidstone
  - Manchester
  - Norwich
  - Oxford
  - Plymouth